## THE EFFECT OF MOTOR IMAGERY TRAINING ON MUSCLE ACTIVITY, MOTOR IMAGERY AND FUNCTIONAL MOVEMENT SKILLS IN INDIVIDUALS UNILATERAL CEREBRAL PALSY

**NCT NUMBER: 03954808** 

**Document Date: 10.06.2020** 

## **Statistical Analysis Plan**

For descriptive statistics, mean and standard deviation or median and minimum-maximum values for numerical variables, number and percentage values for categorical variables were given. Normality assumption was analyzed using the Shapiro Wilks test. Whether there was a difference between the two groups was examined using the significance test of the two means or the Mann-Whitney U test, and whether there was a difference between three or more groups using one-way analysis of variance or the Kruskal Wallis test. Analysis of variance or Friedman test was used in repeated measures to examine whether there was a difference in repeated measurements. Paired comparisons test was used to identify the group/groups that made a difference in cases where there was a difference between groups.

Whether there was a difference between numerical variables was examined using the Pearson or Spearman correlation coefficient. Statistical significance level was p <0.05. Analyzes were performed using IBM SPSS Statistics (Version 21.0. Armonk, NY: IBM Corp.).